CLINICAL TRIAL: NCT04338477
Title: Multizentrische, Offene Studie Zur Beurteilung Der Verträglichkeit Und Wirksamkeit Von Nephrosolid Tabletten Zur Anregung Der Harnausscheidung Bei Probanden/Non-patient Volunteers
Brief Title: Study to Assess Safety and Efficacy of Nephrosolid Tbs to Stimulate Urinary Output in Non-patient Volunteers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: A. Vogel AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 920174
Record Dates: First submitted 2018-01-04; First posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Urine Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nephrosolid (Experimental): Acute dosis day 1: 3X2 Nephrosolid tablets 0.5 h before intake of a meal Long-term dosis days 2-28: 2x1 Nephrosolid tablets 0.5 h before intake of a meal
  Interventions: Drug: Nephrosolid tablets

INTERVENTIONS:
Drug: Nephrosolid tablets — Adminstration of drug

SUMMARY:
Fluid intake and urinary output are measured with /without intake of Nephrosolid tablets in acute ( 1 day application ) and chronic ( 28 days application) therapy.

DETAILED DESCRIPTION:
To evaluate safety and efficacy of Nephrosolid tbs in the stimulation of urinary output in healthy volunteers, all participants in this open-label study will be asked to record their fluid intake and output on day 0 (without study medication), on day 1 (with 3 x 2 tablets study medication, to be taken 1/2 hour before meals) and on day 28 (with 2 x 1 tablets study medication, morning and noon half an hour before meals) and to take 2 x 1 tablet of Nephrosolid on days 2-28. Subjects will complete a diary during the study to record the tablets taken, amount of fluid consumed, weight, physical activity, and urinary measurement. Safety labs (hematology, clinical chemistry) will be performed at each study visit on days -1 and 29.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to record urine volume and fluid consumption over 3 days.
* Written consent to participate in the study.

Exclusion Criteria:

* Disease or comprehension problems (language) that affect the accurate collection and measurement of urine levels over 3 days.
* Taking diuretic drugs, teas, herbal supplements, or systemic corticosteroids.
* Chronic nephropathy (such as glomerulonephritis, analgesic nephropathy, interstitial nephritis).
* Pregnancy or lactation.
* Psychiatric disorders that include suicidality.
* Surgical intervention in the 3 months prior to enrollment or scheduled surgery during the study.
* Known chronic diseases such as dementia, progressive systemic diseases.
* Known alcohol and/or drug addiction.
* Known allergies to goldenrod or birch leaves.
* Participation in one or more other clinical trials in the last 30 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Tolerability as assessed by the treating physician | day 29
  Tolerability is assessed at 2nd visit /study end, after 4 weeks of intake, according to four step scale ( poor, moderate, good, very good)

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Waelti, Dr. med., Principal Investigator
Locations (2):
- Switzerland (2):
  - Privat practice of Dr. med. Bruno Haug, Medizinisches Zentrum Arbon, Arbon, Thurgau
  - Private Practice Dr. med Bernhard Waelti, Freidorf, Thurgau

IPD SHARING:
Plan to Share IPD: No